CLINICAL TRIAL: NCT01429402
Title: Botulinum Toxin to Improve Results in Cleft Lip Repair
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 98-2237C
Record Dates: First submitted 2011-09-04; First posted 2011-09-07 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-08

CONDITIONS: Scar
Keywords: Botulinum toxin A.; Cleft lip scar
MeSH Terms: conditions — Cicatrix | interventions — Botulinum Toxins, Type A; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- study group I (Experimental): For primary lip surgery, immediately after primary lip repair will received botulinum toxin injection (1-2U/kg, at 25U/mL) into the bilateral aberrant oriented orbicularis ocuris muscle via 4 superficial injection site
  Interventions: Drug: Botulinum Toxin Type A
- Study Group II (Experimental): For revision lip surgery, immediately after revision lip surgery 3 injection of 2.5U of botulinum toxin with a distance of 0.5 cm from each injection and operative wound are injected over both sides of upper lip in a adult on the operation room.
  Interventions: Drug: Botulinum Type A
- Control Group I (Placebo Comparator): Similar amount as group I (in C.C.) of normal saline will be injected after primary lip surgery at 3 months of age.
  Interventions: Drug: Normal Saline
- Control II (Placebo Comparator): Similar amount (in C.C.) as Study Group II of normal saline will be injected after revision lip surgery (secondary cleft lip repair).
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Botulinum Toxin Type A — 1-2U/kg, at 25U/mL, into the bilateral aberrant oriented orbicularis ocuris muscle via 4 superficial injection site; only once after surgery. No additional injection is needed
  Other Names: Botox ( Allergan, Inc., Irvine, Calif)
  Arms: study group I
Drug: Botulinum Type A — b. Study group II: For revision lip surgery, immediately after revision lip surgery 3 injection of 2.5U of botulinum toxin with a distance of 0.5 cm from each injection and operative wound are injected over both sides of upper lip in a adult on the operation room just after surgery. (total dosage injected 15U)
  Other Names: Botox ( Allergan, Inc., Irvine, Calif)
  Arms: Study Group II
Drug: Normal Saline — Similar amount (in C.C.) of normal saline as group I will be injected after primary lip surgery at 3 months of age.
  Other Names: NaCl 0.9%
  Arms: Control Group I
Drug: Normal Saline — Similar amount (in C.C.) of normal saline as study group II will be injected after revision lip surgery (secondary cleft lip repair).
  Other Names: NaCl 0.9%
  Arms: Control II

SUMMARY:
Botulinum toxin type A (Botox; Allergan, Inc., Irvine, Calif) is widely used for facial rejuvenation and many other medical indications. It induces chemodenervation through its action on the presynaptic neuron, preventing release of acetylcholine, which leads to functional denervation of striated muscle for 2 to 6 months after injection. The use of botulinum toxin injection to reduce the facial scar is logical because this could reduce the tensile distracting force of the upper lip caused by the orbicularis oris muscle pull. Tollefson has demonstrate that botulinum toxin injection has decrease lip tension after primary lip repair in 3 children at 3-6 months of age The main aim of this randomized trial is to compare whether post-operative peri-surgical-injection of botulinum toxin into bilateral orbicularis oris muscles can improve scar formation for both primary and secondary cleft lip surgery.

DETAILED DESCRIPTION:
This is a randomized controlled trial primarily designed to compare the scarring after primary and secondary cleft lip repair using post-operative botulinum toxin injection. There will be 4 main groups in this study:-

1. Study group I: For primary lip surgery, immediately after primary lip repair will received botulinum toxin injection (1-2U/kg, at 25U/mL) into the bilateral aberrant oriented orbicularis ocuris muscle via 4 superficial injection site (Tollefson TT 2006).
2. Study group II: For revision lip surgery, immediately after revision lip surgery 3 injection of 2.5U of botulinum toxin with a distance of 0.5 cm from each injection and operative wound are injected over both sides of upper lip in a adult on the operation room.
3. Control group I : Similar amount (in C.C.) of normal saline will be injected after primary lip surgery at 3 months of age.
4. Control group II: Similar amount (in C.C.) of normal saline will be injected after revision lip surgery (secondary cleft lip repair).

   4. ELIGIBILITY 4.1 Inclusion criteria for the primary lip repair group (i) Baby born with cleft lip who will receive primary lip repair at 3 months of age (iii) Written informed consent given by parent/guardian.

4.2 Inclusion criteria for the secondary lip repair group (i) Adult > 16 years old. (ii) Moderate to severe secondary cleft lip and/or nose deformity that warrants corrective surgery.

(iii) Written informed consent given by parent/guardian/patient.

4.3 Patient numbers: 60 for primary lip repair and 60 for secondary lip repair

4.31 Sample size calculation: 10 consecutive patient selected from our OPD on march 2009. Vancouver Scar Scale means 4.6 with SD 1.264911 (rage 3-7). If the study group with improvement of 1 is clinical significant, giving power 0.8 with the same SD, the sample size calculated will be 26.

Using Terason Ultrasound (capacity of measured 1/100 cm or 1/10 mm) the scar width mean is 1.13 mm with SD .6201254. If the study group with improvement of 0.5 mm as clinical significant, giving the power of 0.8 with the same SD, the sample size calculated will be 25.

We will use 30 patients for each group.

4.41 Exclusion criteria for primary lip repair

1. Combined other craniofacial anomalies
2. Without permission of parent/guardian, without signed informed consent by parent/guardian.

4.42 Exclusion criteria for the secondary lip repair

1. Less than 15 years old
2. Mild secondary cleft lip and / or nose deformity that does not warrant corrective surgery.
3. Without written informed consent.
4. Without permission of parent/guardian, the patient signed the consent himself.

   5. Botulinum Toxin injection 5.1 For Study group I: Injections are placed into the orbicularis oris muscle 5 mm adjacent to the scar and the vermilion border on each side of the operative wound (A total of 3 injections per side making a total of 6 injections per patient). 1-2U/kg (total dosage for baby) and 2.5 U (adult ) of botulinum toxin (Botox; allergen, Inc., Irvine, Calif) will be used for each injection. A total dosage of 15 U (for adult) will be injected into each patient.

   For control group a similar amount of Normal saline will be injected.

   6. STUDY VISITS AND ASSESSMENTS 6.1 Registration and Randomization (i) Confirmation of eligibility (ii) Information Sheet (iii) Written informed consent (iv) Registration of baby and adult into study and randomization (v) Scheduling of patient for botox injection immediately after surgery.

   6.2 Follow-up Assessments 6.2.1 Vancouver scar scale (Sullivan T 1990) measures pigmentation, vascularity, pliability and scar height on the postoperative 6 month F/U.

   Ultrasonography measurement of the scar (Fong SS 1997)

   For both primary and secondary lip surgery, the patient will receive postoperative follow up during 1wk, 1mo, 3mo, 6mo. On the 1st week postoperative follow up, the stitches will be removed, 3M taping will be placed over the wound to reduce surface tension and minimize the scar formation. On the 6th mo follow up, a lay person will assess the scar using the Vancouver scar and a plastic surgeon will use ultrasonography to measure the scar.

   The Independent T-Student test will be used to analyze the statistical significance between the two groups.

   Photographic measurement of scar The scar width of the patient's picture at 6 month after surgery will be measured using photoshop CS3 extended. One ruler will be placed on the patient's lip before taken the photo. Then the scar width could be measured.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for the primary lip repair group

* Baby born with cleft lip who will receive primary lip repair at 3 months of age
* Written informed consent given by parent/guardian.

Inclusion criteria for the secondary lip repair group

* Adult > 16 years old.
* Moderate to severe secondary cleft lip and/or nose deformity that warrants corrective surgery.
* Written informed consent given by parent/guardian/patient.

Exclusion Criteria:

* Those patient not fit inclusion criteria

Ages: 3 Months to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2000-07; Primary Completion 2010-08 (Actual); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Vancouver Scar scale | 6 month
  Vancouver scar scale measures pigmentation, vascularity, pliability and scar height on the postoperative 6 month F/U.

SECONDARY OUTCOMES:
Ultrasonography scar measurement | 6 month
  On the 6th mo follow up, ultrasonography to measure the scar width will be performed.
Photographic measurement | 6 month
  The scar width of the patient's picture at 6 month after surgery will be measured using photoshop CS3 extended. One ruler will be placed on the patient's lip before taken the photo. Then the scar width could be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Shin Chang, M.D., Principal Investigator — Chang Gung Memorial Hospital; Philip Kuo-Ting Chen, M.D., Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chun Shin Chang, Taoyuan District, Taoyuan, Taiwan

REFERENCES:
- [Background] Tollefson TT, Senders CM, Sykes JM, Byorth PJ. Botulinum toxin to improve results in cleft lip repair. Arch Facial Plast Surg. 2006 May-Jun;8(3):221-2. doi: 10.1001/archfaci.8.3.221. No abstract available. PMID 16702537
- [Background] Gassner HG, Brissett AE, Otley CC, Boahene DK, Boggust AJ, Weaver AL, Sherris DA. Botulinum toxin to improve facial wound healing: A prospective, blinded, placebo-controlled study. Mayo Clin Proc. 2006 Aug;81(8):1023-8. doi: 10.4065/81.8.1023. PMID 16901024
- [Background] Gassner HG, Sherris DA, Friedman O. Botulinum toxin-induced immobilization of lower facial wounds. Arch Facial Plast Surg. 2009 Mar-Apr;11(2):140-2. doi: 10.1001/archfacial.2009.3. No abstract available. PMID 19289689
- [Background] Gassner HG, Sherris DA, Otley CC. Treatment of facial wounds with botulinum toxin A improves cosmetic outcome in primates. Plast Reconstr Surg. 2000 May;105(6):1948-53; discussion 1954-5. doi: 10.1097/00006534-200005000-00005. PMID 10839391
- [Background] Larrabee WF Jr. Treatment of Facial Wounds with Botulinum Toxin A Improves Cosmetic Outcome in Primates. Plast Reconstr Surg. 2000 May;105(6):1954-1955. doi: 10.1097/00006534-200005000-00006. No abstract available. PMID 11242330
- [Background] Lee BJ, Jeong JH, Wang SG, Lee JC, Goh EK, Kim HW. Effect of botulinum toxin type a on a rat surgical wound model. Clin Exp Otorhinolaryngol. 2009 Mar;2(1):20-7. doi: 10.3342/ceo.2009.2.1.20. Epub 2009 Mar 26. PMID 19434287
- [Background] Sherris DA, Gassner HG. Botulinum toxin to minimize facial scarring. Facial Plast Surg. 2002 Feb;18(1):35-9. doi: 10.1055/s-2002-19825. PMID 11823931
- [Background] Wilson AM. Use of botulinum toxin type A to prevent widening of facial scars. Plast Reconstr Surg. 2006 May;117(6):1758-66; discussion 1767-8. doi: 10.1097/01.prs.0000209944.45949.d1. PMID 16651948
- [Derived] Chang CS, Wallace CG, Hsiao YC, Chang CJ, Chen PK. Botulinum toxin to improve results in cleft lip repair: a double-blinded, randomized, vehicle-controlled clinical trial. PLoS One. 2014 Dec 26;9(12):e115690. doi: 10.1371/journal.pone.0115690. eCollection 2014. PMID 25541942
- [Derived] Chang CS, Wallace CG, Hsiao YC, Chang CJ, Chen PK. Botulinum toxin to improve results in cleft lip repair. Plast Reconstr Surg. 2014 Sep;134(3):511-516. doi: 10.1097/PRS.0000000000000416. PMID 25158709